CLINICAL TRIAL: NCT01925105
Title: Comprehensive Geriatric Assessment - Can it Improve Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Anna Engfeldt, MD, Örebro County Council
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFC-162
Record Dates: First submitted 2013-08-13; First posted 2013-08-19 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Quality of Life
Keywords: Polypharmacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optimization of treatment (Experimental): Optimization of treatment of diseases and symptoms
  Interventions: Other: Experimental: Optimization of treatment
- Control (Placebo Comparator): Treatment as usual

INTERVENTIONS:
Other: Experimental: Optimization of treatment — Optimization of treatment of diseases and symptoms
  Arms: Optimization of treatment

SUMMARY:
Like most developed countries the population of Sweden is getting older and consequently the number of individuals with chronic diseases will be an increasing challenge for its healthcare system. To improve care of the frail elderly, wards with a coordinated multidisciplinary team and multidisciplinary mobile teams were established several years ago. Treatment and follow up is planned in accordance to the patients' medical, psychological and functional capabilities (Comprehensive Geriatric Assessment = CGA). There are to our knowledge only few studies concerning CGA applicable to Swedish conditions. We plan to conduct a Swedish study that evaluates if care and treatment with a modified CGA-model in an outpatient setting can improve quality of life for frail older people.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Live in own home
* Reason to believe that the health condition is not optimal or could be optimized
* Meet at least 2/6 of the following criteria: cognitive impairment, general tiredness or dyspnea, have fallen often/afraid to fall, need help with activities of daily living, hospital care ≥3 times within the last 12 months, care problems at home

Exclusion Criteria:

* Psychosis
* Not understand the Swedish language

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Retained or increased quality of life of at least 20% measured by EQ-5D (EuroQOL) after 1 year from baseline. | 1 year from baseline

SECONDARY OUTCOMES:
Readmission to hospital | 1 year from baseline

OTHER OUTCOMES:
The quality of drug treatment | 1 year from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Peter Engfeldt, Professor, Study Chair — Allmänmedicinskt forskningscentrum, AFC, Örebro läns landsting, Box 1613, 70116 Örebro
Locations (1):
- Örebro County Council, Örebro, Örebro County, Sweden